CLINICAL TRIAL: NCT00696449
Title: An Analysis of Adherence and Associated Factors in Subjects Undergoing Differin Gel, 0.1% Treatment of Moderate to Severe Acne Vulgaris
Brief Title: Analysis of Adherence in Subjects Undergoing Differin Gel, 0.1% Treatment of Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00000406; 31219
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Frequent visits (Experimental): This group will be asked to return to the study center on weeks 1, 2, 4 and 8 for office visits (to remind the Subject to apply the study medication); in addition to the study visits on Weeks 6 and 12.
  Interventions: Drug: Adapalene; Behavioral: frequent visits
- Electronic reminder (Experimental): This group will receive a daily electronic reminder by email, text pager, or phone message (approximately at the same time each day) to use the study medication within a 4-hour window after the reminder and will return to the study center for study visits on Weeks 6 and 12.
  Interventions: Drug: Adapalene; Behavioral: electronic reminder
- Parent reminder (Experimental): In this group parents will be prompted by a daily electronic message by email, text pager, or phone message (approximately at the same time each day) to remind the Subject to use the study medication within a 4-hour window after the reminder. Parents will be instructed to then verbally deliver the message to the study Subject. Subjects will return to the study center for study visits on Weeks 6 and 12.
  Interventions: Drug: Adapalene; Behavioral: Parent reminder
- Standard of care (Experimental): This group is considered to be the "standard of care" arm and will return to the study center for study visits on Weeks 6 and 12. This group will not receive any kind of reminders other than the instructions provided by the study staff during the study visits.
  Interventions: Drug: Adapalene; Behavioral: Standard of care

INTERVENTIONS:
Drug: Adapalene — All Subjects will treat the face once daily in the evening.
  Other Names: Differin® Gel, 0.1%
Behavioral: frequent visits — This group will be asked to return to the study center on weeks 1, 2, 4 and 8 for office visits (to remind the Subject to apply the study medication); in addition to the study visits on Weeks 6 and 12.
  Arms: Frequent visits
Behavioral: electronic reminder — This group will receive a daily electronic reminder by email, text pager, or phone message (approximately at the same time each day) to use the study medication within a 4-hour window after the reminder and will return to the study center for study visits on Weeks 6 and 12.
  Arms: Electronic reminder
Behavioral: Parent reminder — In this group parents will be prompted by a daily electronic message by email, text pager, or phone message (approximately at the same time each day) to remind the Subject to use the study medication within a 4-hour window after the reminder. Parents will be instructed to then verbally deliver the message to the study Subject. Subjects will return to the study center for study visits on Weeks 6 and 12.
  Arms: Parent reminder
Behavioral: Standard of care — This group is considered to be the "standard of care" arm and will return to the study center for study visits on Weeks 6 and 12. This group will not receive any kind of reminders other than the instructions provided by the study staff during the study visits.
  Arms: Standard of care

SUMMARY:
The primary objective of this study is to investigate potential differences between four treatment intervention groups in the adherence to treatment with Differin® Gel, 0.1%. Differin is approved by the Food and Drug Administration (FDA) to treat acne.

DETAILED DESCRIPTION:
Subjects will be enrolled and randomized in a 1:1:1:1 ratio to one of four treatment intervention groups. All Subjects will be treated once-daily for 12 weeks with Differin® Gel, 0.1%. The four intervention groups were designated according to follow-up strategies as follows:

* More frequent than normal office visits
* Electronic reminders (voice, e-mail, text messages)
* Parental involvement/intervention reminders
* No intervention or reminders

ELIGIBILITY:
Inclusion Criteria:

* Male or female Subjects of any race, aged 13 to 18 years inclusive,
* Subjects with a diagnosis of moderate to severe Acne vulgaris, measured by lesion counts of a minimum of 15 and a maximum of 50 inflammatory lesions (papules and pustules) on the face, AND a minimum of 30 and a maximum of 125 total lesions. Subjects with nodules may participate in the study.
* Female Subjects of childbearing potential must have a negative urine pregnancy test (UPT).
* Female Subjects of childbearing potential must practice a highly effective method of contraception during the study
* Subjects (and parent/guardian if Subject is under 18 years of age) must be willing and capable of following study instructions to the extent and degree required by the protocol;
* Subjects able to follow study instructions and likely to complete all required visits;
* Subjects/Representative signs the Informed Consent prior to any study procedures. Subjects under the age of 18 must have one parent or guardian read and sign the Informed Assent Form prior to receiving study treatment but the parent(s) or guardian is not required to attend the follow-up visits unless requested;
* Subject must be willing to be photographed and sign a release form allowing photographs to be used.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning a pregnancy during the study,
* Subjects with a condition or who are in a situation which, in the Investigator's opinion, may put the Subject at risk, may confound the study results, or may interfere with the Subject's participation in the study,
* Subjects with known allergy to one of the components of the test products,
* Subjects who have participated in another investigational drug or device research study within 30 days of enrolment, Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), or or severe acne requiring more than topical treatment (e.g. oral isotretinoin);
* Subjects with a beard or other facial hair that might interfere with study assessments;
* Subjects with underlying diseases or other dermatological conditions that require the use of interfering topical or systemic therapy such as, but not limited to, atopic dermatitis, perioral dermatitis or rosacea;
* Subjects who are at risk in terms of precautions, warnings, and contra-indication (see package insert for Differin Gel, 0.1%);
* Subjects who foresee intensive UV exposure during the study (mountain sports, UV radiation, sunbathing, etc.);
* Subjects with a known history of drug and/or alcohol abuse.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Frequent Office Visits: This group will be asked to return to the study center on weeks 1, 2, 4 and 8 for office visits (to remind the Subject to apply the study medication); in addition to the study visits on Weeks 6 and 12.
- Electronic Reminders: This group will receive a daily electronic reminder by email, text pager, or phone message (approximately at the same time each day) to use the study medication within a 4-hour window after the reminder and will return to the study center for study visits on Weeks 6 and 12.
- Parental Reminders: In this group parents will be prompted by a daily electronic message by email, text pager, or phone message (approximately at the same time each day) to remind the Subject to use the study medication within a 4-hour window after the reminder. Parents will be instructed to then verbally deliver the message to the study Subject. Subjects will return to the study center for study visits on Weeks 6 and 12.
- Standard of Care Control: This group is considered to be the "standard of care" arm and will return to the study center for study visits on Weeks 6 and 12. This group will not receive any kind of reminders other than the instructions provided by the study staff during the study visits.
Period: Overall Study
Arm/Group | Frequent Office Visits | Electronic Reminders | Parental Reminders | Standard of Care Control
Started | 15 | 15 | 15 | 16
Completed | 12 | 9 | 14 | 13
Not Completed | 3 | 6 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Frequent Office Visits | Electronic Reminders | Parental Reminders | Standard of Care Control | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 15 | 16 | 61
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 9 | 10 | 34
  Male | 8 | 7 | 6 | 6 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 16 | 61

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Treatment
Description: Percentage of prescribed doses taken over the 12-week study period, as measured by a Medication Event Monitoring System (MEMS) cap
Time Frame: 12 weeks
Measure: Median (Full Range); unit: Percent of prescribed doses
Arm/Group | Frequent Office Visits | Electronic Reminders | Parental Reminders | Standard of Care Control
Number analyzed (Participants) | 15 | 15 | 15 | 16
Percent of prescribed doses | 64 [10 to 98] | 38 [0 to 98] | 28 [5 to 60] | 52 [2 to 83]

ADVERSE EVENTS:
Arm/Group | Frequent Office Visits | Electronic Reminders | Parental Reminders | Standard of Care Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No